CLINICAL TRIAL: NCT01142843
Title: Clinical Preliminary Evidence of the Efficacy of a Mouthwash Containing 5% Propolis for the Control of Plaque and Gingivitis: Phase II Study
Brief Title: Preliminary Evidence of the Efficacy of a Mouthwash Containing 5% Propolis for the Control of Plaque and Gingivitis
Acronym: MGP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Vagner Rodrigues Santos, Universidade Federal de Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSantos-UFMG
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2009-05

CONDITIONS: Dental Plaque; Gingivitis
Keywords: clinical trial; mouthwash; green propolis; dental plaque; gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: green propolis mouthwash — The subjects were instructed to brush their teeth as usual and to rinse with the 10mL of Mouthwash contain 5% Green Propolis, twice a day, for one minute, right after their meals in the morning and at night. The treatment was performed during three months
  Other Names: mouthrinse; Brazilian propolis; Baccharis dracunculifolia

SUMMARY:
Mouthwash based on medicinal plants and propolis can be easily found in the Brazilian market even if it has not been tested in reliable clinical trials on its efficacy or possible unpleasant side effects like the ones which alter the hard and soft oral tissues. The aim of this study was to obtain preliminary evidence of efficacy of an alcohol-free mouthwash containing 5% green propolis (MGP 5%) on the control of plaque and gingivitis. Were chosen twenty-five subjects that are UFMG employees and individuals who would begin treatment on an extension project called Supportive Periodontal Therapy at the Faculty of Dentistry of Federal University of Minas Gerais, Belo Horizonte, from August to December 2009. The subjects went through a dental prophylaxis before starting rinse. They were then instructed to rinse twice a day for a minute, immediately after brushing (morning and night), using the 10 ml of the MGP 5%. After 45 and 90 days using the product the individuals returned for a clinical evaluation which considered changes in the soft and hard oral tissues and involved collecting plaque and gingivitis indexes. On their last appointment the subjects answered a questionnaire about their level of appreciation and acceptability of the mouthwash. Compliance with the treatment was also evaluated through an attendance form. For the statistic analysis we used BioEstat 4.0 and Excel 2007.

DETAILED DESCRIPTION:
The first reference to mouthrinse as a formal practice is credited to Chinese medicine, about 2700 B.C.E., to treatment the diseases of the gums (Fischman, 1997).

The gram-positive and gram-negative bacteria that compose oral biofilms produces many metabolites that induce gingival inflammation (that is, gingivitis). Gingivitis can lead to periodontitis, a condition in which gingival and bone tissues are destroyed. The majority of the population may not perform mechanical plaque removal sufficiently. Thus, antimicrobial mouthrinses that improve daily home care may provide an effective way of removing or controlling bacterial plaque to limit gingivitis and periodontitis (Haffajee et al., 2008).

The main indications are either the improvement of dental health (plaque and gingivitis elimination in particular) or the prevention of infections caused by bacteria of the oral cavity in specific situations, such as tooth extraction, intraoral surgical procedures or immune suppression due to cancer therapy or transplantation. The use of antimicrobial mouthrinses has been proposed to reduce the levels of oral bacteria, specially Streptococcus mutans (Kocak et al., 2009).

In fact, it has been shown that chemotherapeutic mouthrinses are an effective adjunct to regular brushing and flossing for patients with gingivitis, providing a clinically significant benefit in the reduction of plaque and gingivitis (Haffajee et al., 2008).

Propolis is a resinous substance collected by honeybees from buds and exudates of certain trees and plants, and stored inside their hives. It has been used in folk medicine from ancient times to treat various ailments (Kunimasa et al., 2009).

The action against microorganisms is an essential characteristic of propolis, and humans have used it for centuries for its pharmaceutical properties (Kalogeropoulos et al., 2009).

The antibacterial activity of propolis is reported due to flavonoids, aromatic acids and esters present in resins. Galangin, pinocebrin and pinostrobin are known as the flavonoids agents more effective against bacteria. Ferulic acid and caffeic acid also contribute to the bactericidal action of propolis (Marcucci, 1995). Thus, the purpose of this study was to show a preliminary evidence about the effect of an alcohol-free mouthwash containing 5% of green propolis for the control of plaque and gingivitis in subjects for three months.

Materials and Methods

Design study and Product tested

This was an interventional study of phase II for three months, follow up type, and was conducted at the Faculty of Dentistry of Federal University of Minas Gerais, Brazil, from August 2009 to April 2010.

The alcohol-free mouthwash containing 5% green propolis (MGP 5%) used in that study was handled according to our request by PharmaNéctar ® (Belo Horizonte), within the standards required by ANVISA (Brazil, 2000) and within the requirements of ISO 9001 and GMP International (Table 1).

Participants

Twenty five subjects, age varying from 18 to 60 years (median age 35,92 ±9,7), with generally good health, not pregnant nor breastfeeding, who met the following inclusion criteria, were included into the study: a minimum of 20 sound, natural teeth; a mean plaque index (PI) (Turesky modification of the Quigley-Hein Plaque Index, 1970) of at least 1.5; a mean gingival index (GI) (Talbott modification Gingival Index of the Löe-Silness, 1977) of at least 1.0. Subjects with orthodontic appliances or removable prosthetics, tumors of the soft or hard oral tissues, advanced periodontal disease, or that received antibiotic therapy 2 weeks before the start of the study or that presented hipersensibility to propolis were excluded. Third molars and those teeth with cervical restorations or prosthetic crowns were not included in the tooth count. The selection of participants was made by convenience, based especially on the availability for the study, along the study was conducted. All subjects read and signed informed consent forms before the start of the study. The protocol for the study was approved by the local ethical review committee (Committee of Bioethics in Research at the Federal University of Minas Gerais (COEP/UFMG - 0600/09).

Assessing mouthwash

The examination baseline consisted of a complete soft and hard tissues examination that was performed to register the condition of oral mucosa, so that any changes in the course of the study could be identified , making assessment to whether these changes could be related to the mouthrinse. The gingivitis of the mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual, of all elegible teeth was scored using the Talbott modification Gingival Index of the Löe-Silness - GI, 1977, in which the gum was scored on a four-point scale from 0 (absence of inflammation) to 3 ( severe inflammation). The supragingival plaque of the mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual, of all elegible teeth was scored using the Turesky modification of the Quigley-Hein Plaque Index - PI, 1970. Previously, disclosing with erythrosine 3% solution, plaque was scored on a six point scale from 0 (no plaque) to 5 (plaque covers two-thirds or more of the tooth surface). Of the mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual, of all scorable teeth was scored using the Turesky modification of the Quigley-Hein Plaque Index - PI, 1970. There were also evaluated Severity Plaque Index and Severity Gingival Index (Palomo et al., 1989; Volpe et al.,1993). These index measured the rate of the surface that had high count of plaque (count similar to 3, 4, 5 of the modification Quigley-Hein Plaque Index, 1970) and high gingival index (count similar to 2,3 modification Gingival Index of the Löe-Silness, 1977.

These examinations were all repeated after 45 and 90 days of use of mouthrinse. After baseline examination, each subject received a complete oral prophylaxis, which included the removal of all supragingival plaque and calculus deposits. Soon after, the subjects received the 5% green propolis-containing mouthrinse alcohol-free (MGP 5%) and a toothbrush. They were instructed to brush their teeth as usual and to rinse with the 10mL of MGP 5%, twice a day, for one minute, right after their meals in the morning and at night. Participants were required not to use another mouthrinse throughout the study. When new supplies were issued, subjects returned their used materials, so that compliance to theproduct could be monitored.

Reproducibility of clinical examinations

All examinations were conducted by a single examiner trained to optimize the consistency of the study. Prior to the study, the adviser trained the dental examiner, as a "gold standard", directing him to introduce the periodontal probe, gently, into the gingival sulcus,, keeping the instrument parallel to the long axis of the tooth, sliding it from the distal to the mesial so delicately in the buccal and lingual surface of each evaluated tooth. For calibration, there was examined nine subjects not included in the study.

For the plaque index it was performed a theoretical calibration. Soon after, photos were used to obtain a standardization intra-examiner. The photos were exhibited by the adviser to the examiner that noted the values of plaque index corresponding to each picture. After 15 days, the same pictures were exposed to the examiner that noted again the values of plaque index. Next, the plaque index obtained in the first and second time was compared to verify the level of intra-examiner. Then, we obtained a kappa value of 0.73, considered a substantial estimate of reliability (Landis & Koch, 1977).

Statistical Analysis

The statistical package BioEstat version 4.0 was used for data analysis in this study. The average adjusted in the baseline for both scores of the modified Plaque Index of Quigley-Hein (1970) and modified Gingival Index of Löe-Silness (1977) as for the corresponding severity scores, for being a non-parametric distribution, were compared through covariance analysis, by Friedman test for data obtained at 45 and 90 days of the study. All statistical tests of hypotheses had two strands and was considered a significance level of p< 0.05 (Allen et al. 1998; Arweiler et al., 2001).

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* generally good health
* not pregnant nor breastfeeding
* a minimum of 20 sound, natural teeth
* a mean plaque index (PI) (Turesky modification of the Quigley-Hein Plaque Index, 1970) of at least 1.5 or more
* a mean gingival index (GI) (Talbott modification Gingival Index of the Löe-Silness, 1977) of at least 1.0 or more
* signing the terms of agreement

Exclusion Criteria:

* Subjects with orthodontic appliances or removable prosthetics
* Subjects with tumors of the soft or hard oral tissues
* Subjects with advanced periodontal disease
* Subjects that received antibiotic therapy 2 weeks before the start of the study
* Subjects with hipersensibility to propolis confirmed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of a mouthwash containing 5% propolis for the control of gingivitis | 90 days
  Difference in the Gingival Index scores between the start and the end of the study.

SECONDARY OUTCOMES:
Efficacy of a mouthwash containing 5% propolis for the control of plaque | 90 days
  Difference in the Plaque Index scores between the start and the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Minas Gerais (UFMG), Belo Horizonte, Minas Gerais, Brazil